CLINICAL TRIAL: NCT05601817
Title: Virtual Reality and Computerized Cognitive Intervention for Mild Cognitive Impairment in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Miyeon Jung, Assistant Professor, Indiana University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15739; 1K76AG074940-01A1 (NIH)
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Mild Cognitive Impairment
Keywords: heart failure; mild cognitive impairment; older adults; cognitive intervention; cognitive training; attention restoration; virtual reality
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction | interventions — Vitamin A; Mesna

STUDY DESIGN:
Intervention Model Description: A 2 by 2 factorial design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vita (virtual reality-based cognitive restoration intervention) (Experimental): Participants randomized to Vita will receive a virtual reality head-mount device (e.g., Oculus Quest) to view nature pictures for 10 minutes (1 set of 10 pictures)/day, 2-3 days/week for 8 weeks (a total of 20 sets for 200 minutes, approximately 3.3 hours) based on the provided activity schedule. Participants will receive weekly check-in calls from the intervention RA during the 8 weeks of intervention phase.
  Interventions: Behavioral: Vita
- Com (computerized cognitive training intervention ) (Experimental): Participants randomized to Com will receive a tablet computer (e.g., iPad) to complete BrainHQ training for 1 hour (6 exercises)/day, 2-3 days/week for 8 weeks (total of 20 hours) based on the provided activity schedule. Participants will receive weekly check-in calls from the intervention RA during the 8 weeks of intervention phase.
  Interventions: Behavioral: Com
- Vita+Com (Both Vita and Com intervention) (Experimental): Participants randomized to Vita+Com will receive both Vita and Com simultaneously. They will spend 10 minutes on Vita and then 1 hour on Com per day, 2-3 days/week for 8 weeks (a total of 23.3 hours). Participants will receive weekly check-in calls from the intervention RA during the 8 weeks of intervention phase.
  Interventions: Behavioral: Vita+Com
- Usual care (No Intervention): Participants randomized to this control condition will continue to receive their usual care, but no interventions from the study team. We will monitor changes in their activities that may affect changes in cognitive function (e.g., starting book clubs) by weekly check-in calls during the 8 weeks of intervention phase.

INTERVENTIONS:
Behavioral: Vita — Vita is developed by this study team based on Attention Restoration Theory. The Vita intervention involves viewing 360 degree nature pictures on a virtual reality headset.
  Arms: Vita (virtual reality-based cognitive restoration intervention)
Behavioral: Com — Com intervention uses BrainHQ from PositScience that was developed based on the brain neuroplasticity. The com intervention involves doing game-like training on a iPad.
  Arms: Com (computerized cognitive training intervention )
Behavioral: Vita+Com — Vita+Com intervention is a combination of both Vita and Com interventions. Participants will be asked to complete Vita first and then Com intervention.
  Arms: Vita+Com (Both Vita and Com intervention)

SUMMARY:
This research project is relevant to public health because both heart failure (HF) and mild cognitive impairment (e.g., trouble remembering and concentrating beyond normal aging) are highly prevalent among older adults in the United States. Despite advances in health care, there are no effective interventions for treating cognitive impairment in HF, which if left untreated, leads to suboptimal health, quality of life, and shorter survival. Therefore, the investigators propose to test the effect of a dual-component intervention comprised of a virtual reality-based cognitive restoration intervention and computerized cognitive training on cognitive function and overall health among 172 older adults with HF who experience mild cognitive impairment.

DETAILED DESCRIPTION:
Heart failure (HF) and mild cognitive impairment (MCI) are prevalent among older adults in the U.S. Patients with HF are twice as likely to have MCI than people without HF. Cognitive impairment in HF is associated with significant decline in one's ability to take care of one's self and higher 12-month mortality. A small number of cognitive interventions have demonstrated preliminary efficacy in improving cognitive function in HF. However, this work suffers from some major limitations: 1) lack of focus on patients who already have cognitive impairments and at higher risk of dementia; 2) focus on single-component interventions; 3) lack of evaluation of responsiveness variables including genetic biomarkers; and 4) lack of long-term follow-up. Dr. Miyeon Jung, PhD, RN proposes to address this gap by conducting a randomized controlled pilot trial to estimate the preliminary efficacy of a virtual reality-based cognitive restoration (Vita) combined with a computerized cognitive training intervention (Com) relative to each intervention alone and standard of care among 172 older HF patients with MCI. The Specific aims of the project are to estimate the effects of the Vita and Com interventions individually and in combination to improve: 1) attention and memory (Aim 1); 2) HF self-care, instrumental activities of daily living, and health-related quality of life (Aim 2); and 3) dementia free survival (Aim 3) over 1 year. An exploratory aim is to examine moderating factors that may influence intervention efficacy (i.e., baseline cognitive function, depressive symptoms, HF severity, and presence of apolipoprotein E ε4 and BDNF Met allele).

ELIGIBILITY:
We will use a two-step process to screen and enroll the patients. First, we will screen potentially eligible patients from the Indiana University Health systems using these eligibility criteria.

Inclusion Criteria:

1. ≥ 55 years;
2. chronic HF Stage C validated from echocardiography or comparable measure or B-type natriuretic peptide (BNP) level > 400 pg/ml [or equivalent NT-proBNP] in past 3 years;
3. ability to communicate in English;
4. capacity to consent according to the Indiana University Institutional Review Board policies, or lacks capacity to consent but has the ability to provide assent from someone who can serve as LAR; and
5. Subjectively reported cognitive concern assessed by the question, "Do you have any trouble with your memory or thinking?".

Exclusion Criteria:

1. pre-HF (Stages A and B) or advanced HF (Stage D);
2. vision or hearing problems that can interfere with cognitive testing;
3. major neurological disorder (e.g., previously diagnosed dementia, Parkinson's disease, epilepsy, multiple sclerosis);
4. major psychiatric disease (e.g., schizophrenia, bipolar disorder);
5. life-threatening unstable illness other than HF (e.g., end-stage cancer); and
6. users of regular computerized cognitive training or participants in cognitive training trials in the past year.

Second, we will enroll patients only if they have MCI or normal cognition by not meeting criteria for dementia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive function: attention | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Trail Making and Number Span Test from National Alzheimer's Coordinating Center Neuropsychological battery (Uniform Data Set V3.0)
Changes in cognitive function: memory | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Craft Story 21 and Benson Figure Copy for memory from National Alzheimer's Coordinating Center Neuropsychological battery (Uniform Data Set V3.0)

SECONDARY OUTCOMES:
Changes in heart failure self-care | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Self-Care of Heart Failure Index
Changes in instrumental activities of daily living | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Functional Activities Questionnaire (for both patients and informants)
Changes in instrumental activities of daily living | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Everyday Problems Test (performance-based, for patient only)
Changes in health-related quality of life | Baseline, 8 weeks, 16 weeks, and 1 year (52 weeks) after baseline
  Minnesota Living with Heart Failure Questionnaire
Dementia-free survival | 1 year after baseline
  Survival status (alive or deceased) at year collected from electronic health records

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided